CLINICAL TRIAL: NCT01206088
Title: A Phase IV Study for Nilotinib in Patients With Imatinib-resistant or Intolerant Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia (CML) in Chronic or Accelerated Phase.
Brief Title: Tasigna in Glivec-resistant or Intolerant Patients in CML
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107AKR02
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: CML; Nilotinib; Imatinib Resistant; Imatinib Intolerant
MeSH Terms: interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nilotinib (Experimental)
  Interventions: Drug: nilotinib

INTERVENTIONS:
Drug: nilotinib — administration of nilotinib as 2nd line

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of nilotinib in patients with Imatinib resistant or intolerant CML-CP or AC. Efficacy evaluation will be made by Complete cytogenetic response rate(CCyR) at 12 months after nilotinib administration.

ELIGIBILITY:
Inclusion Criteria:

* Imatinib resistant chronic myelogenous leukemia in chronic phase with cytogenetic confirmation of Philadelphia chromosome.
* Documented chronic phase CML as defined by:

  * < 15% blasts in peripheral blood and bone marrow
  * < 30% blasts plus promyelocytes in peripheral blood and bone marrow
  * < 20% basophils in the peripheral blood
  * ≥ 100 x 109/L (≥ 100,000 /mm3) platelets
  * No evidence of extramedullary leukemic involvement, with the exception of hepatosplenomegaly
  * the patients with no CHR(complete hematologic response) after 3 months treatment, no mimical cytogenetic response(Ph+<65%) after 6 months treatment, no major cytogenetic response(Ph+<35%) after 12 months treatment.

Or

* Imatinib resistant Philadelphia positive CML-AC will be defined as at lease one following and no bast crisis before treatment.

  * <30% and ≥ 15% blasts in peripheral blood and bone marrow
  * ≥ 30% blasts plus promyelocytes in peripheral blood and bone marrow
  * ≥ 20% basophils in the peripheral blood
  * < 100 x 109/L (≥ 100,000 /mm3) platelets without related treatment
  * progression of CML-AP with Imatinib treatment, no hematologic response in bone marrow after at least 4 weeks treatment with imatinib. Progression from AP will be defined by increased numbers more than 50% of peripheral WBCs, blasts, basophils and platelets.
* definition of Imatinib intolerance in CML-CP and AP

  * the patients who discontinued imatinib treatment with any dosage due to Grade 3 or 4 non-hematologic adverse event or Grade 4 hematologic adverse event sustained for more than 7 days even best complementary therapy.
* WHO performance scale ≤ 2
* provide signed informed consent form

Exclusion Criteria:

* Cardiac dysfunction : LVEF <45% by echocardiography, using pacemaker,Congenital long QT syndrome or a known family history of long QT syndrome, History of or presence of clinically significant ventricular or atrial tachyarrhythmias, Clinically significant resting brachycardia (<50 beats per minute),QTc > 450 msec on baseline ECG (using the QTcF formula), Myocardial infarction within 12 months prior to starting study, Other clinically significant heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension).
* Known cytopathologically confirmed CNS infiltration (in absence of suspicion of CNS involvement, lumbar puncture not required).
* Severe or uncontrolled medical conditions (i.e. uncontrolled diabetes, active or uncontrolled infection).
* History of significant congenital or acquired bleeding disorder unrelated to cancer.
* Treatment with any CSGF within 1 week of Day 1 except Erythropoietin.
* History of non-compliance to medical regimens or inability to grant consent.
* Use of therapeutic coumarin derivatives (i.e., warfarin, acenocoumarol, phenprocoumon)
* Patients with another primary malignancy except if the other primary malignancy is neither currently clinically significant or requiring active intervention
* Patients actively receiving therapy with strong CYP3A4 inhibitors (e.g, erythromycin, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir, mibefradil) and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug. See link for complete list of these medications: http://medicine.iupui.edu/flockhart/table.htm.. Novartis must be contacted if a patient needs to be started on any of these drugs during study treatment.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery)
* History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis.
* patients who diagnosed HIV infection.
* patients who has hypersensitivity for nilotinib or its additives
* Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug (Please see http://www.torsades.org/medical-pros/drug-lists/printable-drug-list.cfm for a comprehensive list of agents that prolong the QT interval)
* Patients who are: (a) pregnant, (b) breast feeding, (c) of childbearing potential without a negative pregnancy test prior to baseline and (d) male or female of childbearing potential unwilling to use contraceptive precautions throughout the trial
* Patients with rare genetic disease such as galactose intolerance, moderate lactase deficiency or glucose-galactose absorption disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2009-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Complete cytogenetic response (CCyR) rate | at 12 months

SECONDARY OUTCOMES:
evaluation of safety by NCI-CTCAE version 3.0 | until 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- St. Mary hospital, Catholic medical center, Seoul, South Korea